CLINICAL TRIAL: NCT04041934
Title: Effect of the Quality of Dietary Proteins on the Sleep Young Elite Athletes and the Obese Adolescent
Acronym: Protmorpheus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RBHP 2018 FANTINI; 2018-A02680-55 (Other: 2018-A02680-55)
Record Dates: First submitted 2019-04-05; First posted 2019-08-01 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Obese Adolescent; Elite Adolescent Athletes
Keywords: sleep; adolescent; tryptophan; athletes; obeses
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Intervention Model Description: Tryptophan (Trp) / Large neutral amino acids (Lnaa) ratio of proteins taken varies-double-blind between sessions
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cohorte 1 (Experimental): Tryptophan (Trp) / Large neutral amino acids (Lnaa) ratio = 0.11
  Interventions: Dietary Supplement: tryptophan
- cohorte 2 (Experimental): Tryptophan (Trp) / Large neutral amino acids (Lnaa) ratio = 0.07
  Interventions: Dietary Supplement: tryptophan
- cohort 3 (Experimental): Tryptophan (Trp) / Large neutral amino acids (Lnaa) ratio = 0.04
  Interventions: Dietary Supplement: tryptophan

INTERVENTIONS:
Dietary Supplement: tryptophan — Each experimental session will be carried out over a week. Adolescents will take part randomly in three sessions. In order to limit inter-individual differences, the diet of the first 3 days will be fixed to the RDA followed by 3 days where dietary intake will be supplemented with different protein (PROT REF : ratio = 0,04 PROT1 : ratio = 0,07, session PROT2 : ratio = 0,11). Tryptophan (Trp) / Large neutral amino acids (Lnaa) ratio of proteins taken varies-double-blind between sessions. All proteins had the same dose and packages. Neither the researcher nor the participants were aware of the quality of the protein.

SUMMARY:
Adolescence is characterized by major transitions in sleep and circadian rhythm. This rapid pivotal period increases the risks of sleep debt and poor sleep quality, leading to pronounced diurnal fatigue and drowsiness . Some adolescent's populations are more vulnerable than others to poor sleep. Obesity and elite sports involvement are two factors that have been distinctly associated with disturbed sleep. Several studies show that obesity was associated with a decrease in sleep efficiency and increased arousals . On the other hand, recent studies point out that sleep problem is widespread in young athletes which substantially increase the risks of injury, burnout and concussions .

Despite the importance of sleep in holistic development, physical (i.e. recovery, metabolism, muscle growth, weight control), cognitive (i.e. learning, memory, decision-making, Vigilance) and athletic performances (Fullagar et al., 2015).

A wide range of recent papers emphasize that some nutrients take part in the regulation of internal clock and sleep quality. The effect of tryptophan (Trp) on sleep was lifted on the basis of the serotonergic hypothesis. Serotonin (5-HT) is synthesized from Trp circulating in the brain following two-step procedure in raphe neurons. Serotonin, in turn, is a precursor of melatonin and both molecules contribute to the regulation of sleep-wake behaviors. However, Trp is an essential amino acid, which means that it cannot be synthesized by the organism, and must exclusively be provided via degradation of proteins from the diet. The passage of tryptophan to the brain is assured through carrier disposed at the blood-brain barrier level. However, carrier transport depends on other competitive amino acids (LNAAs: leucine, isoleucine, valine, phenylalanine, and tyrosine). Therefore, increased brain uptake of tryptophan does not depend only on Trp concentrations but rather on the blood Trp / LNAA ratio.

PROTMORPHEUS trial, was designed to examine how supplementation with proteins of different Trp/LNAA ratio affect sleep on adolescents (obese, athletes) with mild sleep disturbances.

DETAILED DESCRIPTION:
Double-blind controlled pre-post trial where each subject acts as his own control.

Three measurement sessions will be performed for each teenager. Each session will be conducted over a week. Each teenager will participate in three protein enrichment sessions: PROT1 session, PROT2 session, and Tryptophan ratio (Trp) / neutral amino acids (AAN) reference session (PROT REF) (PROT1: ratio = 0.07, PROT2 session: ratio = 0.11 and PROT REF session: ratio = 0.04). During these sessions the protein intake will be doubled with regard to recommended dietary intakes through the consumption of protein shakes (from 0.8 g per kg of body weight to 1.6 g per kg).

At each session:

* 2 EEG sleep assessments
* 2 evaluations of the biological profile from fasting blood samples
* 2 evaluations of melatonin peak from salivary specimens
* 1 assessment of physical activity and sedentary lifestyle
* 1 evaluation of the metabolic response to submaximal exercise
* 1 assessment of muscle strength and fatigue
* 1 assessment of cognitive performance Control of food intake (3 days at RDI + 3 days with doubled protein intake) will be achieved by preparing meals and weighing food. An evaluation of the ad libitum food intake of the 7th day will be carried out by the weighing method.

  1. peripheral quantitative computed tomography (pQCT) of the muscular cross-section (thigh and forearm) at the beginning of the study

ELIGIBILITY:
Inclusion Criteria:

* young athletes OR adolescent with BMI > 90 percentiles

Exclusion Criteria:

* Disorders and / or pathology of sleep and chronic diseases of the digestive tract
* Medical or surgical history not compatible with the study, any other chronic illness or injury that may interfere with the subject's abilities
* Take medication that may interfere with the results of the study (corticosteroids ...) or sleeping pills
* Surgical intervention in the previous 3 months
* Regular consumption of tobacco, cannabis or alcohol
* Special diet

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Change effect of a supplementation with proteins of different Trp/Lnaa ratio on sleep of elite adolescent athletes with mild sleep disturbances | Change from pre-intervention
  Efficiency of sleep (ratio of time spent in bed / sleep time)

SECONDARY OUTCOMES:
change in biochemical marker related to sleep | day4 day7
  measured by blood test : GH, GHRH, TSH, Sérotonine (5HT), Kynurénine, Tryptophane
Change in biochemical markers related food intake | day4 day7
  measured by blood test : Insuline, Leptine, Ghreline, Adiponectine, GLP-1, PYY3-36, Nesfatine, Irisine
change in biochemical markers related to inflammation | day4 day7
  measured blood test : CRP-us, IL1b, IL6, TNF-alpha, IL4, IL10, sTNFR1 and sTNFR2
Resting metabolic rate kcal per day | day 7
  Resting metabolic rate. Resting metabolic rate (RMR) will be measured under fasted state, using indirect calorimetry (MetaMax 3b, Cortex Biophysik, Leipzig, Germany). In agreement with the manufacturer's recommendations gas analysis will be calibrated before the test. The test will be held in a thermoneutral environment (22-25 °C). Participants will extend in a supine position for 45 min before starting the measurements. After achieving a steady state, O2 consumption and CO2 production standardized for temperature, barometric pressure and humidity will be recorded at 1 min intervals for 20-45 min and will be averaged over the whole measurement period. After that, RMR (in kcal/day) and respiratory quotient (ratio of CO2/O2) will be calculated.
muscular fatigue | day 7
  force measurement : Time in second spent on 60% of MVIC (Maximal Voluntary Isometric Contraction (MVIC) of the knee flexors)
Cognitive performances | day 7
  Measures by cognitive tests : Stroop test
Cognitive performances | day 7
  Measures by cognitive tests :Trail marking test
Cognitive performances | day 7
  Measures by cognitive tests : Barrage test
Cognitive performances | day 7
  Measures by cognitive tests : PASAT
Cognitive performances | day 7
  Measures by cognitive tests : Symbol digit test
Energy intake | day 7
  Energy intake and proportion of the energy derived from each class of macronutrient (carbohydrate, fat, and protein) measured on meals offered "ad-libitum"

CONTACTS AND LOCATIONS:
Overall Officials: Livia Fantini, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France